CLINICAL TRIAL: NCT01002365
Title: Perioperative Hyperoxygenation and Wound Site Infection Following Surgery for Acute Appendicitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Other Study IDs: Bickel10-2009
Record Dates: First submitted 2009-10-25; First posted 2009-10-27 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Acute Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Post op care (Active Comparator)
  Interventions: Other: Oxygen delivery; Other: Oxygen administration
- Oxygen administration- different % (Active Comparator)
  Interventions: Other: Oxygen administration

INTERVENTIONS:
Other: Oxygen delivery
  Arms: Post op care
Other: Oxygen administration

SUMMARY:
Patients undergoing open appendectomy for acute appendicitis were enrolled in a randomized prospective study.

ELIGIBILITY:
Inclusion Criteria:

* Consent was given
* 15 years old or older
* Underwent acute appendicitis

Exclusion Criteria:

* Lack of follow up
* Younger than 15 years
* Not eligible according to physician decision

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Western Galilee Hospital, Nahariya, Israel

REFERENCES:
- [Derived] Bickel A, Gurevits M, Vamos R, Ivry S, Eitan A. Perioperative hyperoxygenation and wound site infection following surgery for acute appendicitis: a randomized, prospective, controlled trial. Arch Surg. 2011 Apr;146(4):464-70. doi: 10.1001/archsurg.2011.65. PMID 21502457